CLINICAL TRIAL: NCT02001259
Title: Efficacy of Epidural Steroid in Controlling Postoperative Pain After Primary Total Knee Arthroplasty: A Randomized Double-blinded Controlled Trial
Brief Title: Efficacy of Epidural Steroid for Controlling Pain After Primary TKA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Thammasat University (Other)
Responsible Party: Principal Investigator, Supakit Kanitnate, orthopaedic department, Thammasat University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: orthoTU05
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: Postoperative Pain
Keywords: post-operative pain control; total knee arthroplasty; epidural steroid injection
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Epidural lidocaine (Active Comparator): epidural lidocaine: 3 mL of 1% lidocaine with adrenaline and 3 mL of 1% lidocaine without adrenaline into epidural catheter at 48 hr after surgery
  Interventions: Drug: epidural lidocaine
- epidural triamsinolone (Experimental): epidural triamsinolone: 40 mg of triamsinolone (1 mL), 2.5 mL of 1% lidocaine with adrenaline and 2.5 mL of 1% lidocaine without adrenaline into epidural catheter at 48 hr after surgery
  Interventions: Drug: epidural triamsinolone

INTERVENTIONS:
Drug: epidural triamsinolone — add drugs into catheter at 48 hr after surgery
  Other Names: epidural steroid
  Arms: epidural triamsinolone
Drug: epidural lidocaine — add into catheter at 48 hr after surgery
  Other Names: epidural xylocaine
  Arms: Epidural lidocaine

SUMMARY:
The purpose of this study is to determine efficacy of epidural steroid for postoperative pain control after TKA

DETAILED DESCRIPTION:
Epidural triamsinolone can reduce postoperative pain and longer duration of pain control after TKA

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis of the knee who undergoing unilateral primary total knee arthroplasty
* 50-85 years old
* ASA class 1-3

Exclusion Criteria:

* unable to perform epidural anaesthesia
* history of drug allergies: lidocaine, steroid
* renal impairment (CrCl <30 mL/min)
* liver impairment
* cognitive function disorders
* displacement of epidural catheter

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
post-operative pain | 3 months
  measured with VAS for pain (VAS at rest and on motion)

SECONDARY OUTCOMES:
functional knee score | 3 months
  measured with WOMAC

OTHER OUTCOMES:
complication of epidural triamcinolone | 2 weeks
range of motion of the knee | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Supakit Kanitnate, M.D., Principal Investigator — orthopaedic department
Locations (1):
- department of orthopaedic surgery, Faculty of medicine, Thammasat university, Khlong Luang, Changwat Pathum Thani, Thailand